CLINICAL TRIAL: NCT06020690
Title: A Clinical Study to Evaluate the Safety and Effectiveness of Novabel Bioabsorbable Steroid-releasing Stent for the Chronic Sinusitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Enlight Medical Technologies (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YM-2023-003
Record Dates: First submitted 2023-08-15; First posted 2023-09-01 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Chronic Sinusitis
Keywords: bioabsorbable; steroid-releasing stent

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novabel bioabsorbable steroid-releasing stent (Experimental)
  Interventions: Device: bioabsorbable steroid-releasing stent
- marketed bioabsorbable steroid-releasing stent (Active Comparator)
  Interventions: Device: bioabsorbable steroid-releasing stent

INTERVENTIONS:
Device: bioabsorbable steroid-releasing stent — The patient after functional endoscopic sinus surgery to treat their chronic sinusitis, the experimental device or active comparator device will be implanted to the sinus to prevent re-intervention (surgery or medicine).
  Other Names: functional endoscopic sinus surgery

SUMMARY:
The goal of this clinical trial is to learn about the safety and effectiveness of Novabel bioabsorbable steroid-releasing stent in chronic sinusitis. The main questions it aims to answer are:

* The safety of this device for the chronic sinusitis
* The effectiveness of this device for the chronic sinusitis Participants will be implanted bioabsorbable steroid-releasing stents after FESS surgery. Participants will be asked to be back to the clinic for follow-up 14 days, 30 days, 90 days, 180 days and 360 days after procedure.

Researchers will compare test device and marketed device to see if the safety and effectiveness between these two devices are non-inferior.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose with CRS based on Chinese guidelines for diagnosis and treatment of chronic rhinosinusitis (2018), who were scheduled to undergo primary or revision bilateral ESS.
* Have evidence of bilateral sinus based on computed tomographic (CT) scan (Lund-Mackay [L-M] score of <=3 on each side).
* Can understand the purpose of this study and will to join and finish all the follow up according to the study. Sign the ICF.

Exclusion Criteria:

1. Know history of allergy or intolerance to corticosteroids or mometasone furoate.
2. The subject has a known allergic reaction or contraindication to the device material and its degradation products (L-polylactic acid, racemic polylactic acid, lactide lactate, lactic acid).
3. Clinical evidence of cystic fibrosis, severe polyposis or sinonasal tumors.
4. Clinical evidence of acute bacterial sinusitis or suspicion of invasive fungal sinusitis.
5. Glaucoma, ocular hypertension, posterior subcapsular cataracts.
6. Known history of immune deficiency or concurrent condition requiring active chemotherapy and/or immunotherapy management for the disease.
7. Clinical evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments during the 360 day follow-up period.
8. Current ESS including frontal sinus surgery is aborted for any reason.
9. Pregnant or lactating female
10. Investigator determination that the potential study subject is unable to comply with study procedures and/or follow-up, or provided informed consent.
11. Currently involved in another clinical study where that participation may conflict or interfere with the treatment, follow-up or results of the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-09-09 (Estimated); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
non reintervention rate | 30 days
  The need for postoperative interventions, medical and surgical, as determined based on review of video endoscopic findings by an independent blinded surgeon.

SECONDARY OUTCOMES:
Lund-Kennedy score | 30 days, 90 days, 180 days and 1 year
  Lund-Kennedy endoscopic scoring system based on polyps, oedema, discharge, scarring and crusting. from 0-2 is None/absent; mild; severe.
Lund-Mackay score | 90 days
  Each side of sinus is graded separately: 0 (no abnormality); 1 (partial opacification); 2 (complete opacification). If there is no frontal sinus (aplasia), the score is 0. Scores were calculated based on the results of a paranasal sinus CT scan 1-3 mm axial slice thickness with coronal and sagittal reconstruction. Result: score 0-24.
VAS score | 30 days, 90 days, 180 days and 1 year
  A 100mm VAS, ranging from 0 (no pain) to 100 (very severe pain), is used to measure pain intensity throughout the previous 24h.
sinus panty rate | 30 days, 90 days, 180 days and 1 year
  as determined based on review of video endoscopic findings by an independent blinded surgeon
implantation successful rate | immediately after the procedure

OTHER OUTCOMES:
adverse event rate | immediately after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Li, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, China